CLINICAL TRIAL: NCT04534270
Title: Efficacy and Safety of Dapagliflozin in Non-diabetic Children With Proteinuria
Brief Title: Efficacy and Safety of Dapagliflozin in Children With Proteinuria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Hong Xu，MD.PhD, Professer, Children's Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EASODICWP.01
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-02

CONDITIONS: Proteinuria
Keywords: proteinuria; SGLT2i
MeSH Terms: conditions — Proteinuria | interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dapagliflozin treatment (Experimental)
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin will be given 5mg per day (weight≤30kg) or 10mg per day (weight>30kg), for 12 weeks

SUMMARY:
The purpose of the study is to investigate the antiproteinuric effect of Dapagliflozin in children with proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 years to 18 years;
* Urinary protein excretion > 0.2g in a 24-hr urine collection;
* eGFR≥60 ml/min/1.73m2;
* No history of diabetes;
* On stable doses of ACE inhibitors or angiotensin receptor blockers (ARBs) for > 1 month;

Exclusion Criteria:

* Receiving immunosuppressive therapy within three months prior to enrolment.
* Blood pressure less than 5th percentile of the same gender, age, and height -
* Leukocyte and/or nitrite positive urinalysis that is untreated;
* History of organ transplantation, cancer, liver disease;
* Evidence of hepatic disease as determined by any one of the following: ALT or AST values exceeding 3x ULN at the screening visit;
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
The change in 24-hr proteinuria after a 4 weeks treatment with dapagliflozin | From baseline to weeks 4
  Urine will be collected for 24 hours and total urinary protein will be detected

SECONDARY OUTCOMES:
The change in 24-hr proteinuria after a 12 weeks treatment with dapagliflozin | From baseline to weeks 12
  Urine will be collected for 24 hours and total urinary protein will be detected
The change in eGFR after a 12 weeks treatment with dapagliflozin | Measured at baseline, weeks 4, weeks 8, weeks 12
  eGFR are repeated measurement data and will be evaluated by Schwartz formula（k*height（cm)/creatinine(umol/L), k=36.5）

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China